CLINICAL TRIAL: NCT05725395
Title: Virtual Reality Education for Hospitalized Pediatric Patients Improves Intrinsic Motivation: A Prospective Crossover Study
Brief Title: Virtual Reality as a Intrinsic Motivation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Caruso (Other)
Responsible Party: Sponsor-Investigator, Thomas Caruso, Clinical Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 68166
Record Dates: First submitted 2022-11-22; First posted 2023-02-13 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Psychological
Keywords: Virtual Reality
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality then Standard of Care (Experimental): Participants will be randomized to receive the virtual reality intervention on the first day and receive standard of care on the second day of in-patient care.
  Interventions: Behavioral: Virtual Reality; Behavioral: Standard of Care
- Standard of Care then Virtual Reality (Experimental): Participants will be randomized to receive the standard of care on the first day and receive virtual reality intervention on the second day of in-patient care.
  Interventions: Behavioral: Virtual Reality; Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Virtual Reality — During in-patient care participants will be randomized to receive or not receive the educational virtual reality intervention on the first day. After two days, participants will receive a total of 10 minutes interventional in the morning (between 8am to 12pm) every day until their in-patient care concludes.
Behavioral: Standard of Care — For case control, participants will service as their self control and be randomized to receive no virtual reality intervention on either the first day or the second day of in-patient care.

SUMMARY:
The goal is to explore the use of Virtual Reality (VR) as an intervention to increase intrinsic motivation in a healthcare setting. The investigators would like to determine if an educational VR intervention in the course of healthcare could increase pediatric patient intrinsic motivation compared to standard of care (i.e no VR).

DETAILED DESCRIPTION:
While virtual reality has gained momentum as a therapeutic supplement to distract from pain perception and to reduce anxiety, it has received less attention as an intervention to promote more holistic psychological intrinsic motivation in the course of in-patient care. Child and adolescent self-reported measures of intrinsic motivation have also been looked over in favor of parent or practitioner measures of a child's intrinsic motivation.

To evaluate the effectiveness of virtual reality on child and adolescent intrinsic motivation while undergoing hospital care, the investigators will determine the effect of virtual reality to 1) increase pediatric patient intrinsic motivation compared to standard of care using educational virtual reality, 2) establish a comprehensive profile of short-term psychological well-being in school-aged children and adolescents following admission to a hospital. Participants will serve as their own control to either receive intervention on the first day or second day of the in-patient care and no intervention will be given on the other day.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age range from 5 to 25 at LPCH/SHC facilities
* patient who speak english only

Exclusion Criteria:

* Participants who do not consent
* Have a history of seizure disorder
* Currently have nausea
* Have motion sickness
* Are clinically unstable
* Currently using corrective glasses (not compatible with VR headset)
* Currently pregnant
* non-English speakers

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 158 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in the intrinsic motivation | Day 1(baseline), Day 2
  Measured with six items from the modified Intrinsic Motivation Inventory (IMI) - Interest/Enjoyment Subscale. The perceived interest/enjoyment is scored on scale ranging from 1 (Not at all true) to 7 (very true)

SECONDARY OUTCOMES:
Change in current mental well being as measured by the modified WHO (Five) Well-Being Index | Day 1(baseline), Day 2
  The modified WHO (Five) Well-Being Index is a participant-reported outcome measure that assesses current mental well being. Questionnaire contains 5 questions . Scores range from 0 to 5, with higher scores indicating the corresponding feeling exists all the time.
Change in the self-esteem (child) | Day 1(baseline), Day 2
  Measured with five items from the modified Rosenberg Self-Esteem Scale (child). The self-esteem is scored on scale ranging from 1 (very true) to 4 (Definitely not true)
Change in the self-esteem (Adolescent) | Day 1(baseline), Day 2
  Measured with five items from the modified Rosenberg Self-Esteem Scale (Adolescent). The self-esteem is scored on scale ranging from 1 (Strongly agree) to 4 (Strongly disagree)
Change in the caregiver perception of the educational experience of the patient | Day 1(baseline), Day 2
  Measured with seven items from a modified Educational Experience Parental Survey Scale. The caregiver perception of the educational experience of the patient is scored on scale ranging from 1 (strongly disagree) to 7 (strongly agree)
Change in educational self efficacy | Day 1(baseline), Day 2
  Measured with six items from the modified New General Self-Efficacy Scale. The educational self efficacy is scored on scale ranging from 1 (strongly disagree) to 5 (strongly agree)

OTHER OUTCOMES:
Change in the Positive and Negative Affect feeling and emotion for Children | Day 1(baseline), Day 2
  Measured with ten items from the Positive and Negative Affect Schedule for Children (PANAS-C). The positive affect (PA) and negative affect (NA) feelings and emotions are scored on scale ranging from 1 (Very slightly or not at all) to 5 (Extremely)

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Kern ML, Benson L, Steinberg EA, Steinberg L. The EPOCH Measure of Adolescent Well-Being. Psychol Assess. 2016 May;28(5):586-97. doi: 10.1037/pas0000201. Epub 2015 Aug 24. PMID 26302102
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Duckworth AL, Peterson C, Matthews MD, Kelly DR. Grit: perseverance and passion for long-term goals. J Pers Soc Psychol. 2007 Jun;92(6):1087-101. doi: 10.1037/0022-3514.92.6.1087. PMID 17547490
- [Background] Duckworth AL, Quinn PD. Development and validation of the short grit scale (grit-s). J Pers Assess. 2009 Mar;91(2):166-74. doi: 10.1080/00223890802634290. PMID 19205937
- [Background] Rosenberg M. [Consciousness from the viewpoint of electrophysics]. Psychiatr Neurol Med Psychol (Leipz). 1965 Nov;17(11):408-10. No abstract available. German. PMID 5884740
- [Background] Lachman ME, Weaver SL. The sense of control as a moderator of social class differences in health and well-being. J Pers Soc Psychol. 1998 Mar;74(3):763-73. doi: 10.1037//0022-3514.74.3.763. PMID 9523418
- [Background] Kallem S, Carroll-Scott A, Rosenthal L, Chen E, Peters SM, McCaslin C, Ickovics JR. Shift-and-persist: a protective factor for elevated BMI among low-socioeconomic-status children. Obesity (Silver Spring). 2013 Sep;21(9):1759-63. doi: 10.1002/oby.20195. Epub 2013 May 13. PMID 23671041